CLINICAL TRIAL: NCT06926816
Title: Universal Genetic Testing for Cancer Risk Reduction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 23-00413
Record Dates: First submitted 2025-04-11; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Genetic Testing
Keywords: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Completed genetic screening test (Experimental): Participants will complete point-of-care genetic testing by saliva test. Participants with actionable pathogenic variants will be referred to the appropriate specialists to discuss risk-reduction strategies and offered genetic counseling. All Participants will be given the opportunity for genetic counseling, and if interested and desired this will be facilitated by the research team.
  Interventions: Genetic: Natera® Empower™ hereditary cancer panel test; Other: Specialist Referral
- Denied genetic screening test (No Intervention): Participants in this arm have declined the genetic screening test.

INTERVENTIONS:
Genetic: Natera® Empower™ hereditary cancer panel test — The test will be the Natera® Empower™ hereditary cancer panel test and will be collected by saliva.
  Arms: Completed genetic screening test
Other: Specialist Referral — Participants with actionable pathogenic variants will be referred to the appropriate specialists (e.g., medical oncologist, gynecologic oncologist, breast surgeon) to discuss risk-reduction strategies and offered genetic counseling
  Arms: Completed genetic screening test

SUMMARY:
The purpose of this research study is to see if offering genetic testing for cancer-related genes is feasible and acceptable for patients presenting for gynecology clinic visits, instead of needing to see specialized providers or needing to meet specific criteria. The primary aim to assess the proportion of patients who undergo genetic testing, and the proportion of patients with pathogenic variants.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients between ages of 25-39 years at the time of visit
2. Receive gynecologic care at an affiliated NYU Langone Health (NYULH) site listed in this protocol.

Exclusion Criteria:

1. Personal history of ovarian, fallopian tube, primary peritoneal, or uterine cancers
2. Previously undergone germline testing for ovarian cancer risk variants (prior commercial saliva-based kits, such as 23andMe, are acceptable)
3. History of bilateral salpingo-oophorectomy
4. Visit related to pregnancy or immediately postpartum (within 2 weeks)

Ages: 25 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who undergo genetic testing | Up to 9 months
  Outcome measure will be assessed via review of electronic medical record (EMR).

SECONDARY OUTCOMES:
Number of participants with pathogenic variants | Up to 9 months
  Outcome measure will be assessed via review of Natera® Empower™ hereditary cancer panel test results.

CONTACTS AND LOCATIONS:
Overall Officials: Bhavana Pothuri, MD, MS, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: bhavana.pothuri@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to bhavana.pothuri@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.